CLINICAL TRIAL: NCT03601130
Title: Post Market Clinical Follow up - Assessment of HydroxyColl Bone Graft Substitute in High Tibial Osteotomy Wedge Grafting.
Brief Title: Assessment of HydroxyColl Bone Graft Substitute in High Tibial Osteotomy Wedge Grafting.
Acronym: HColl_HTO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: SurgaColl Technologies Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SC100.2
Record Dates: First submitted 2018-07-03; First posted 2018-07-26 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Osteoarthritis, Knee
Keywords: osteotomy; osteoarthritis; bone graft substitute
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No Bone Graft (Other): Open Wedge High Tibial Osteotomy with medial plate fixation (without bone grafting)
  Interventions: Device: DePuy Synthes TomoFix Medial High Tibial Plate (MHT) fixation (Standard of Care)
- HydroxyColl Bone Graft Substitute (Active Comparator): Open Wedge High Tibial Osteotomy with medial plate fixation (with bone grafting) using Hydroxycoll bone graft substitute.
  Interventions: Device: HydroxyColl Bone Graft Substitute; Device: DePuy Synthes TomoFix Medial High Tibial Plate (MHT) fixation (Standard of Care)

INTERVENTIONS:
Device: HydroxyColl Bone Graft Substitute — The intervention involves the use of Open Wedge High Tibial Osteotomy with DePuy Synthes TomoFix Medial High Tibial Plate (MHT) fixation (Standard of Care) with the HydroxyColl bone graft substitute i.e. bone graft substitute vs. no bone graft substitute.
  Arms: HydroxyColl Bone Graft Substitute
Device: DePuy Synthes TomoFix Medial High Tibial Plate (MHT) fixation (Standard of Care) — The intervention involves the use of Open Wedge High Tibial Osteotomy with DePuy Synthes TomoFix Medial High Tibial Plate (MHT) fixation (Standard of Care) without the HydroxyColl bone graft substitute i.e. bone graft substitute vs. no bone graft substitute.

SUMMARY:
The overall goal of this study is to demonstrate the safety and efficacy of Hydroxycoll bone graft substitute when used in the treatment of patients undergoing surgical treatment for varus mis-alignment in medial unicompartmental osteoarthritis of the knee. HydroxyColl bone graft substitute will be evaluated when utilized in Open Wedge High Tibial Osteotomy with medial plate fixation. Its safety profile will be evaluated as defined by the number of reported adverse events.

DETAILED DESCRIPTION:
Osteoarthritis (OA) of the knee is joint damage, resulting in pain accompanied by varying degrees of functional limitation and reduced quality of life. 20% of adults over 50 and 40% over 80 years report disability from knee pain secondary to osteoarthritis.The majority of patients present to primary care with symptoms of pain and stiffness, which reduces mobility and with associated reduction in quality of life, with many patients not requiring surgery, with their symptoms adequately controlled by non-surgical measures. When patient's symptoms are not controlled by up to 3 months of non-operative treatment they become candidates for assessment for joint surgery. There are a number of surgical (Arthroscopy, Total/Partial Knee Replacement, High Tibial Osteotomy) and non-surgical (including exercise, weight loss, manual therapy, oral medication, injection therapy, splints and braces) options available. The decision to undergo surgery is based on patient symptom pattern, with the type of surgery determined by the pattern of joint damage and the patient's preference. High Tibial Osteotomy (HTO) should be considered primarily for patients with varus mis-alignment in medial unicompartmental osteoarthritis of the knee as the main indication for the procedure. HTO involves removing or adding bone to realign the limb and offload the knee. It is effective and can provide functional outcomes similar to those seen after joint replacement. HTO is a commonly used surgical procedure and has wide appeal because of the preservation of the knee joint. The principal advantages of opening wedge high tibial osteotomy include maintenance of the bone stock, correction of the deformity close to its origin, and no requirement for a fibular osteotomy. Although it is a good option for young patients with isolated medial compartment OA and varus deformity, it can be done even for older active people over 65. By preserving the patient's own knee anatomy, a successful osteotomy may delay the need for a joint replacement for several years. Another advantage is that there are no restrictions on physical activities after an osteotomy, even high impact exercise.

Contemporary Surgical approaches to HTO can often utilise bone graft substitutes to improve patient outcomes. Bone grafting in open wedge high tibial osteotomy (HTO) is an area of clinical research that requires further evaluation. While open wedge high tibial osteotomy (OWHTO) with medial plate fixation is a proven adequate and safe method for treatment of medial compartment osteoarthritis of the knee and varus deformity, particularly in young and/or active, it nevertheless creates a gap in the metaphysis of the tibia. To enhance bone healing and increase initial mechanical stability, a high degree HTO may require the application of bone graft/substitute to fill the osteotomy gap. Moreover, HTO has been associated with risk of nonunion, collapse and loss of correction. Autologous bone graft is the "gold standard" to fill the bone defect, but iliac crest graft harvest has risks. The associated complications include pain, thigh hypoesthesia, infection, pelvic bone fracture and discomfort wearing clothes. Allograft is commonly used to avoid the risks of autografting, such as donor side morbidity. However, the use of allograft increases additional risks such as disease transmission, immunologic reactions and slow remodelling. Due to the limited autologous bone availability and the problem of donor-site morbidity, many efforts have been made to find adequate supporting material for augmentation after osteotomy. Hydroxyapatite, β-tricalcium phosphate or the combination of both are the most commonly used synthetic augments in HTO. However, the most suitable material for filling the opening space in OWHTO has not been conclusively identified. While HTO with and without bone grafting has been assessed as radiologically equivalent, of particular interest to clinicians and patients is the contention around the secondary outcomes (site morbidity and bleeding, chronic pain, patient discomfort long term) which are frequently a challenge in postoperative management of patients. Autologous bone graft would still be the best choice for a lot of applications where bone grafting is needed but there are many disadvantages - the relatively high donor morbidity and the limited amount which can be harvested - which will eventually lead to a very restricted use of it. Allografts do not have these limitations, but in the form of demineralized bone matrix they have very variable osteoinductive properties and can possibly transmit diseases. Synthetic 2nd generation biomaterials have a long and safe history of use but do not provide a compelling alternative to traditional bone grafting. 3rd generation biomaterials as bone graft substitutes, such as HydroxyColl, offer exciting prospects of improved patient clinical outcomes and may provide a viable alternative to autologous bone grafts. Treatment for these patients would be with Open Wedge High Tibial Osteotomy with medial plate fixation. Over the period of the trial, adverse events will be reported by the study centre and it will be the prominence or absence of these, along with blood inflammatory marker evaluations that will determine the inherent safety of Hydroxycoll compared to the standard of care. At each follow up visit x-rays will be performed and evaluated by a certified radiologist. Site morbidity and bleeding will be clinically assessed. They will report and assess the radiographic images determining if healing has occurred. Along with the clinical assessment, the surgeon or a member of the clinical team will determine extent of healing. Patients will also self-report a number of key pain, mobility and post-operative joint inflammation outcomes.

The study is a single centre randomized blinded study to assess the efficacy and safety of Hydroxycoll bone graft substitute used as a bone graft substitute in Open Wedge High Tibial Osteotomy with DePuy Synthes TomoFix Medial High Tibial Plate (MHT) fixation (Standard of Care). This study has been designed to last for 52 weeks with follow up visits post surgery, 6 weeks, 12 weeks and a final follow-up at 52 weeks. In case of AEs/SAEs ongoing when the patient has completed the study, the patient will be contacted by phone one month after study completion for follow-up. The study will have 2 arms with 20 subjects per arm, each receiving at the time of surgical intervention either; 1) Open Wedge High Tibial Osteotomy with medial plate fixation (without bone grafting). 2) Open Wedge High Tibial Osteotomy with medial plate fixation (with bone grafting) using Hydroxycoll bone graft substitute. An Independent Review Board (IRB) will approve the protocol before the study begins. A clinical monitor selected by SurgaColl will monitor the trial. Any serious adverse events (SAE) will be reported as soon as possible (within 48 hours of awareness) to SurgaColl by the study centre. SurgaColl will communicate the SAE to all relevant authorities.

ELIGIBILITY:
Inclusion Criteria:

* Able to give written informed consent to participate in this study
* Both male and females who will be admitted to the hospital for treatment of varus mis-alignment in medial unicompartmental osteoarthritis of the knee of the degree to which the surgeon deems it necessary to include a bone grafting procedure
* Kellgren-Lawrence grade 1-4
* Ability and willingness to comply with all study requirements

Exclusion Criteria:

* History or presence of the following conditions: known sensitivity to bovine collagen or hydroxyapatite materials; diabetes, immune-compromised, vascular disease, metabolic/systemic bone disorder, osteomyelitis
* Failure to provide written informed consent
* Severe acute or chronic medical illness, including symptomatic cardiovascular disease
* Weight less than 40 kilograms
* Any clinically significant abnormality at the time of submission, in the judgement of the investigator would preclude safe completion of the study
* Any use of estrogens, estrogen-progestin therapy, selective estrogens receptor modulators (SERMs) or calcitonin within 3 months, and use of bisphosphonates or recombinant PTH 1-34, 1-84 or other PTH fragments/analogues within the last 6 months
* History of alcohol or drug abuse within the last year
* History of non-compliance to medical regimens and/or patients who are considered potentially unreliable
* Significant psychiatric disorder or behaviour
* Presence of any concomitant condition which, in the opinion of the investigator or the sponsor, may interfere with the interpretation of efficacy and safety data gathered in this study including chronic infections
* Chronic or >7 days concomitant use of oral corticosteroids within 1 month prior to screening
* Regular smoker (more than 10 cigarettes per day) for the last 12 months
* Participation in another interventional orthopaedic clinical trial within 1 month of the beginning of this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-04-30 (Actual); Primary Completion 2019-12-27 (Estimated); Study Completion 2020-04-29 (Estimated)

PRIMARY OUTCOMES:
Radiological Healing | Week 6
  clinical assessment of healing based on radiological observations by a member of the clinical team
Radiological Healing | Week 12
  clinical assessment of healing based on radiological observations by a member of the clinical team
Radiological Healing | Week 52
  clinical assessment of healing based on radiological observations by a member of the clinical team
Knee injury and Osteoarthritis Outcome Score (KOOS) | Day 0
  Patient reported outcomes relating to knee pain and function (Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL)). KOOS consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL). Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
Knee injury and Osteoarthritis Outcome Score (KOOS) | Day 1
  Patient reported outcomes relating to knee pain and function (Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL)). KOOS consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL). Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
Knee injury and Osteoarthritis Outcome Score (KOOS) | Week 6
  Patient reported outcomes relating to knee pain and function (Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL)). KOOS consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL). Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
Knee injury and Osteoarthritis Outcome Score (KOOS) | Week 12
  Patient reported outcomes relating to knee pain and function (Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL)). KOOS consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL). Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
Knee injury and Osteoarthritis Outcome Score (KOOS) | Week 52
  Patient reported outcomes relating to knee pain and function (Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL)). KOOS consists of 5 subscales; Pain, other Symptoms, Function in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL). Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
EQ5D Score | Day 0
  Patient reported outcomes relating to mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels (1-5): no problems, slight problems, moderate problems, severe problems and extreme problems.
EQ5D Score | Day 1
  Patient reported outcomes relating to mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels (1-5): no problems, slight problems, moderate problems, severe problems and extreme problems.
EQ5D Score | Week 6
  Patient reported outcomes relating to mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels (1-5): no problems, slight problems, moderate problems, severe problems and extreme problems.
EQ5D Score | Week 12
  Patient reported outcomes relating to mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels (1-5): no problems, slight problems, moderate problems, severe problems and extreme problems.
EQ5D Score | Week 52
  Patient reported outcomes relating to mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels (1-5): no problems, slight problems, moderate problems, severe problems and extreme problems.
VAS Score | Day 0
  Patient reported outcomes relating to pain. Visual analog scale [VAS] is a measure of pain intensity. It is a continuous scale comprised of a horizontal (called horizontal visual analogue scale) or,vertical called vertical visual analog scale usually 10 cm or 100 mm length [both the gradations are used]. It is anchored by two verbal descriptors, one for each symptom extreme.For pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [on 100-mm scale].
VAS Score | Day 1
  Patient reported outcomes relating to pain. Visual analog scale [VAS] is a measure of pain intensity. It is a continuous scale comprised of a horizontal (called horizontal visual analogue scale) or,vertical called vertical visual analog scale usually 10 cm or 100 mm length [both the gradations are used]. It is anchored by two verbal descriptors, one for each symptom extreme.For pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [on 100-mm scale].
VAS Score | Week 6
  Patient reported outcomes relating to pain. Visual analog scale [VAS] is a measure of pain intensity. It is a continuous scale comprised of a horizontal (called horizontal visual analogue scale) or,vertical called vertical visual analog scale usually 10 cm or 100 mm length [both the gradations are used]. It is anchored by two verbal descriptors, one for each symptom extreme.For pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [on 100-mm scale].
VAS Score | Week 12
  Patient reported outcomes relating to pain. Visual analog scale [VAS] is a measure of pain intensity. It is a continuous scale comprised of a horizontal (called horizontal visual analogue scale) or,vertical called vertical visual analog scale usually 10 cm or 100 mm length [both the gradations are used]. It is anchored by two verbal descriptors, one for each symptom extreme.For pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [on 100-mm scale].
VAS Score | Week 52
  Patient reported outcomes relating to pain. Visual analog scale [VAS] is a measure of pain intensity. It is a continuous scale comprised of a horizontal (called horizontal visual analogue scale) or,vertical called vertical visual analog scale usually 10 cm or 100 mm length [both the gradations are used]. It is anchored by two verbal descriptors, one for each symptom extreme.For pain intensity, the scale is most commonly anchored by "no pain" (score of 0) and "pain as bad as it could be" or "worst imaginable pain" (score of 100 [on 100-mm scale].

SECONDARY OUTCOMES:
Safety outcome based on clinical assessment of the adverse events reported during the trial. | Day 0
  Safety outcome based on clinical assessment of the adverse events reported during the trial specifically related to the Hydroxycoll and compared to standard of care.
Safety outcome based on clinical assessment of the adverse events reported during the trial | Day 1
  Safety outcome based on clinical assessment of the adverse events reported during the trial specifically related to the Hydroxycoll and compared to standard of care.
Safety outcome based on clinical assessment of the adverse events reported during the trial | Week 6
  Safety outcome based on clinical assessment of the adverse events reported during the trial specifically related to the Hydroxycoll and compared to standard of care.
Safety outcome based on clinical assessment of the adverse events reported during the trial | Week 12
  Safety outcome based on clinical assessment of the adverse events reported during the trial specifically related to the Hydroxycoll and compared to standard of care.
Safety outcome based on clinical assessment of the adverse events reported during the trial | Week 52
  Safety outcome based on clinical assessment of the adverse events reported during the trial specifically related to the Hydroxycoll and compared to standard of care.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Risebury, MA MBBS FRCS, Principal Investigator — Hampshire Hospitals NHS Foundation Trust
Locations (1):
- Basingstoke & North Hampshire Hospital, Basingstoke, United Kingdom